CLINICAL TRIAL: NCT07174765
Title: Population-Based Analysis of Incidence and Mortality of Septic Shock: The Registry of Administrative Data Automatically Recorded-Septic Shock Project
Brief Title: Population-Based Analysis of Incidence and Mortality of Septic Shock
Acronym: RADAR
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital de Granollers (Other)
Responsible Party: Principal Investigator, Josep M Badia, Prof, Hospital de Granollers
Other Study IDs: RADAR-Septic Shock Project
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Septic Shock
Keywords: Sepsis; Septic shock
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Association; Comorbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a diagnosis of septic shock: All patients with a diagnosis of septic shock discharged hospitals of the public hospital network of Catalonia, Spain, were included.
  Interventions: Other: Person-level linkage of the database looking for relationship with septic shock survival and comorbidities, previous intake of medication, and previous dependence on health services.

INTERVENTIONS:
Other: Person-level linkage of the database looking for relationship with septic shock survival and comorbidities, previous intake of medication, and previous dependence on health services. — A descriptive analysis of the baseline demographics, risk factors, health status, comorbidities, frailty, and previous dependence on health services of all patients admitted with septic shock to hospitals in the region will be carried out.
  The overall data of patients admitted to hospitals will be analysed. The survival data of patients will be compared with their previous individual drug consumption and inhospital survival to septic shock. In addition, drug dependence and dependence on health services of survivors will be studied in comparison with their situation prior to sepsis.
  The objective is to establish the Registry of Administrative Data Automatically Recorded for Septic Shock (RADAR-Septic Shock), leveraging administrative data to characterize septic shock incidence, describe patient profiles, identify population-specific healthcare needs, and provide benchmark values for performance assessment in Catalonia's public health system.

SUMMARY:
RADAR-Septic Shock is a population-based observational study in Catalonia (Spain) that will identify all hospital discharges with septic shock between 2018 and 2023 using an audited population-based registry. The project will quantify incidence, describe patient characteristics and resource use, and compare risk-adjusted in-hospital mortality across hospitals to support quality improvement. Cases are defined by ICD-10 codes for septic shock (R65.21) and post-procedural septic shock (T81.12XA). In preliminary cohort counts, >31,000 episodes were identified across 2018-2023; in 2023 the incidence was ~78 per 100,000 inhabitants with an overall in-hospital mortality of ~33%, higher in hospital-acquired than community-acquired episodes

DETAILED DESCRIPTION:
Septic shock is the most severe manifestation of sepsis and remains a leading cause of death and healthcare utilisation. Outcomes vary by patient mix (age, comorbidities), acquisition setting, infection source, and hospital performance, underscoring the need for robust, population-level surveillance to guide policy and care pathways. RADAR-Septic Shock leverages routinely collected administrative data to provide standardised measures of incidence, resource use, and outcomes across an entire regional health system.

The study aims to quantify the population incidence of septic shock and describe patient demographics, comorbidity burden, infection sources, organ failures, and use of life-support therapies; 2) estimate in-hospital and short-term mortality and length of stay; and 3) benchmark hospitals using risk-adjusted observed-to-expected (O/E) mortality to identify variation and inform improvement strategies.

It is a population-based cohort using the Catalan Minimum Basic Data Set for Acute Care Hospitals (CMBD-HA), an audited, mandatory discharge registry covering all acute-care hospitals in the public system. The analytic period spans January 2018-December 2023.

It will include all hospital discharges containing a primary or secondary diagnosis code for septic shock (ICD-10-CM R65.21) or post-procedural septic shock (T81.12XA). This definition prioritises specificity and uniformity across centres. Episodes will be stratified by acquisition setting (community- vs hospital-acquired).

Extracted variables include: demographics (age, sex); comorbidities and morbidity burden (Adjusted Morbidity Groups [GMA] index); infection source; organ failures; advanced life-support interventions (mechanical ventilation, renal replacement therapy, ECMO); ICU admission; length of stay; and mortality.

Primary outcome: in-hospital mortality. Secondary outcomes: 30-day mortality (where available), ICU admission, length of stay, and use of life-support therapies. Preliminary registry summaries show >31,000 episodes across 2018-2023 and, for 2023, an incidence of ~78 per 100,000 with in-hospital mortality ~33% overall (higher in hospital-acquired episodes). These figures motivate the benchmarking component.

Descriptive statistics will summarise case mix and care processes, including incidence rates per 100,000 inhabitants. Multivariable logistic regression will estimate individual mortality risk; model performance will be assessed (e.g., AUROC) and used to generate expected mortality for each hospital. Comparative performance will be reported via O/E mortality ratios with confidence intervals. Length of stay will be modelled after appropriate transformation. Sensitivity analyses will explore the impact of acquisition setting, infection source, organ failures, and comorbidity burden.

Based on audited counts, the registry includes 31,480 septic shock episodes over 2018-2023 (6,182 in 2023), ensuring sufficient precision for risk modelling and hospital-level benchmarking across the regional network.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of septic shock admitted to the hospitals of the public hospital network of Catalonia, Spain. Septic shock will be defined using the methodology described by Angus et al., which is currently referenced for population-based studies, consisting of coding a diagnosis of infection with acute organ failure, or sepsis or septic shock.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of septic shockadmitted to the hospitals of the public hospital network of Catalonia, Spain, will be included. The data will be obtained from the Catalan Health System (CatSalut) Minimum Basic Data Set (CMBD) registers (compulsory admissions register for all public and private acute care hospitals in Catalonia, Spain, over a 6-year period (2018 and 2023).
Sampling Method: Non-Probability Sample
Enrollment: 31480 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Death due to septic shock | From date of hospital admission until the date of hospital discharge, assessed up to 12 months
  Inhospital death after an episode of septic shock requiring hospital or ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Badia, MD, PhD, Study Director — Hospital General de Granollers
Locations (1):
- Hospital General de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Restrictions apply to the availability of these data, which belong to a national database and is not publicly available.